CLINICAL TRIAL: NCT05121129
Title: Treatment of Major Depression by Magnetic Stimulation Repeated Transcranial on Prefrontal Cortex: Study of Underlying Mechanisms
Brief Title: Treatment of Major Depression by rTMS on Dorsolateral Prefrontal Cortex: Study of Underlying Mechanisms
Acronym: DEPSTIM
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Collaborators: Fondation de France (Other); iBRAIN (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020/477
Record Dates: First submitted 2021-10-13; First posted 2021-11-16 (Actual); Last update posted 2022-12-19 (Actual); Status verified 2022-12

CONDITIONS: Depressive Disorder, Major
Keywords: depression; iTBS; neuronal mechanism; MRI; EEG
MeSH Terms: conditions — Depressive Disorder, Major; Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- iTBS (Experimental): Subjects suffering of MDD assigned to start the trial by 25 sessions of iTBS applied in left DLPFC
  Interventions: Device: iTBS

INTERVENTIONS:
Device: iTBS — 25 active iTBS sessions (5 sessions of 9.5 minutes/day, 1,800 pulses per session, 90% of resting motor threshold, placed over the left DLPFC)

SUMMARY:
The study aims to evaluate the impact of repeated Transcranial Magnetic Stimulation (rTMS) on underlying neuronal mechanisms of adults suffering from major depression disorder (MDD). Short- and long-term effects are assessed by High-Resolution electroencephalography (HR-EEG) or Magnetic Resonance Imaging (MRI) records, experimental tasks and self-rated scales.

DETAILED DESCRIPTION:
Depression is associated with functional and structural changes in the brain, notably in DLPFC (DorsoLateral PreFrontal Cortex). High-frequency rTMS (10 Hz) applied to the left DLPFC is associated with a response rate 3.75 times and remission 2.52 higher than placebo for the treatment of MDD with more reproducible results than those observed for the others rTMS stimulation modalities (low frequency, iTBS5). rTMS is validated as an indication for the treatment of MDD by all learned societies and regulatory authorities in a large number of countries, except in France. Limiting factors concern the lack of knowledge of the action mechanisms, due in particular to the absence of studies based on animal models, the focused application of TMS in rodents being a challenge that few teams have mastered. The rationale for the therapeutic use in the treatment of MDD is now based on some functional brain imaging data showing that rTMS induces a lasting change in brain activity at the site of stimulation (CPFDL) but also in remote interconnected areas such as the limbic region or the amygdala. The DEPSTIM clinical project is part of a translational project with a fundamental approach in rodents.

The main objective is to demonstrate that remission following rTMS of CPFDL occurs via the activation of CPFDL projections to these dysfunctional subcortical areas in MDD.

With a prospective, open design, this study aims to evaluate the impact of iTBS over the left DLPFC on neuronal mechanisms of adults suffering from MDD. Subjects will be submitted to 25 intermittent TBS (iTBS) stimulation sessions for five consecutive days (5 sessions of 9.5 minutes/day, 1,800 pulses per session, 90% of resting motor threshold, placed over the left DLPFC, as mentionned by Cole et al, 2018 (Stanford Neuromodulation Therapy: SNT)). Baseline measures will be compared to those obtained immediately after the end of sessions (Day 5 (D5): short-term effects with HR-EEG analysis), and 30 days (D30) later (long-term effects with MRI analysis).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of MDD (Diagnostic and Statistical Manual of Mental Disorders V [DSM-V] and (Mini International Neuropsychiatric Interview [MINI] criteria, QIDS-C16≥18)
* Right-handed
* No response at a first antidepressant
* Under AD ≥ 6 weeks
* No contraindications for rTMS and MRI
* Absence of addictive comorbidities
* Absence of severe progressive neurologic and/or somatic pathologies (specially tumors, neurodegenerative diseases)
* Inpatients or outpatients of Adult Psychiatric Department
* Signed informed consent form
* Subjects affiliated to or beneficiary from a French social security regime

Exclusion Criteria:

* Subjects under 35 years old or over 65 years old
* Treated with over 4 AD for the current episode
* ECT or rTMS for current episode
* BZD or antiepileptic (except pregabalin up to 75 mg / d, zopiclone ≤7.5 mg / d)
* Left-handed
* Subject under measure of protection or guardianship of justice
* Presence of psychiatric comorbidities
* Subject beneficiary from a legal protection regime
* Subject unlikely to cooperate or low cooperation stated by investigator
* Subject not covered by social security
* Pregnant woman
* Subject being in the exclusion period of another study or provided for by the "National Volunteer File

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-10-13 (Actual); Primary Completion 2023-03-09 (Estimated); Study Completion 2023-04-09 (Estimated)

PRIMARY OUTCOMES:
Change from baseline connectivity with theta wave on EEG at D5 (immediate effect) : | baseline (Day 0), Day 5 post-treatment
  changes in brain connectivity will be analyzed with theta wave
Change from baseline connectivity with beta wave in EEG at D5 (immediate effect) | baseline (Day 0), Day 5 post-treatment
  changes in brain connectivity will be analyzed with beta wave
Change from baseline connectivity with P3 wave EEG at D5 (immediate effect) | baseline (Day 0), Day 5 post-treatment
  changes in brain connectivity will be analyzed with P3 wave
Change from baseline connectivity with fMRI at D30 (prolonged effect) : Resting State Magnetic Resonance Imaging (MRI) | baseline (Day 0), Day 30 post-treatment
  Resting State MRI will allow us to investigate the functional connectivity in the brain, by looking at resting state networks

SECONDARY OUTCOMES:
Severity of depressive symptoms evaluated by the clinician | baseline (Day 0), Day 5 (end of iTBS sessions), Day 12 and Day 30 post-iTBS
  Score achieved on the validated clinician questionnaire Quick Inventory of Depressive Symptomatology (QIDS-C16) evaluating the severity of depressive symptoms.
  The QIDS-C16 was derived from specified items in the IDS-C30, clinician-rated scale to assess the severity of a participant's depressive symptoms. Total scores range from 0-27, with a score of 0 indicating no depression and a score of 27 indicating the most severe depression. Negative change from baseline values indicate improvement in the severity of depression.
Severity of depressive symptoms evaluated by the patient | baseline (Day 0), Day 5 (end of iTBS sessions), Day 12 and Day 30 post-iTBS
  Score achieved on the validated self-reported (QIDS-SR16) evaluating the severity of depressive symptoms. QIDS-SR-16 is a standard questionnaire "The Quick Inventory of Depressive Symptomatology" (16-Item) (Self-Report). This covers questions on falling asleep, sleep during the night, waking up , sleeping too much, feeling sad ,appetite, weight, concentration , how they view themselves, thoughts of death and suicide, general interests, energy levels, feeling slowed down , feeling restless.
Impulsivity | baseline (Day 0), Day 5 (end of iTBS sessions), Day 12 and Day 30 post-iTBS
  Score achieved on the validated Barratt Impulsiveness Scale (BIS-10) evaluating impulsivity. The French version of the BIS-10 is a self-rated 34 item questionnaire, composed by three subscales: motor-impulsivity, cognitive-impulsivity and non-planning-impulsivity. Each item is scored on a 0 to 4 points scale. Higher scores indicate higher levels of impulsivity.
Average adjusted pump scores on the Balloon Analogue Risk Task (BART) | baseline (Day 0), Day 12 post-iTBS
  In the BART participants blow up a series of virtual balloons. With each pump: (a) they earn 5 cents that accumulate in a temporary reserve, but (b) the likelihood of the balloon exploding increases. When this occurs participants lose the money in their temporary reserve. At any time, participants can choose to transfer their earnings to a permanent savings bank (and move to the next balloon). Thus, participants weigh the likelihood of the negative outcome (i.e., the balloon exploding and losing money) with the potential gains (i.e., 5 cents per pump). In the low ambiguity version of the task, the likelihood of the balloon exploding is known. In the high ambiguity version, the likelihood of the balloon exploding is unknown. The average adjusted pump score = average number of pumps on trials in which the balloons did not explode.
Delay Discounting | baseline (Day 0), Day 5 (end of iTBS sessions), Day 12 and Day 30 post-iTBS
  Score achieved on the validated MCQ scale (Monetary Choice Questionnaire), assessing delay discounting. Participants will be asked to make a series of hypothetical choices between small, sooner (impulsive) vs. larger, later (self controlled) hypothetical monetary outcomes
Dimensions of personality | baseline (Day 0), Day 5 (end of iTBS sessions), Day 12 and Day 30 post-iTBS
  Based on the Five-Factor Model, personality traits will be assessed by the French Big Five Inventory questionnaire (BFI-Fr). The BFI-Fr contains 45 self-descriptive statements that assess the 5 personality traits: neuroticism (which refers to a propensity to experience negative emotions, distress, and anxiety), extraversion (a propensity to be energetic, sociable, and experience positive emotions); openness to experience (the tendency to be curious, imaginative, and to entertain new ideas, values, and experiences); conscientiousness (reflecting self-disciplined, planful, and organized); and agreeableness (which refers to cooperativeness and altruism). Each item was rated on a 5-point Likert scale ranging from 1 (strongly disagree) to 5 (strongly agree). All items will be recoded in the direction of the trait label, and the mean will be taken across items for each personality trait.
Motivation | baseline (Day 0), Day 12 post-iTBS
  Score achieved on the validated EEfRT (Effort Expenditure for Rewards Task as an Objective Measure of Motivation and Anhedonia) experimental task. A measure of effort-based decision-making in humans, the Effort Expenditure for Reward Task (EEfRT), will be used. The EEfRT requires participants to choose between a low-effort, low reward task vs a high-effort, high reward task. Willingness to exert effort, or reward motivation, is measured by taking the average number of hard task choices from the first 50 trials.
Social exclusion | baseline (Day 0), Day 12 post-iTBS
  Score achieved on the validated CyberBall experimental task: a ball tossing playing game in which the experimentor can control the number of throws received by the participants. The task is into 2 parts : first, inclusion condition (Participating in wich they will receive 33% of the throw : 10 in a total of 30) and second, exclusion condition (Participating in wich they will receive 2 time the ball in the 10 first throw then none of them in the last 20 throw).
Cognitive assessment | baseline (Day 0), Day 30 post-iTBS
  neuropsychological assessments included in Rapid battery tests (Bereau et al., 2015)
To assess the optimal b-value (a key parameter) for DTI (Diffusion Tensor Imaging) | baseline (Day 0), Day 30 post-iTBS
  b-value is a key technique parameter for DTI, which will decide the quality of DTI image.
  DTI is a sensitive probe of cellular structure that works by measuring the diffusion of water molecules. The measured quantity is the diffusion coefficient, a proportionality constant that relates diffusive flux to a concentration gradient and has units of mm2/s.
C-Reactive Protein (CRP) concentrations | baseline (Day 0), Day 12 post-iTBS
  C-reactive protein rate
Serum Interleukin-6 (IL-6) level | baseline (Day 0), Day 12 post-iTBS
  the measurement of serum IL-6 level in blood
Smoking (tobacco addiction) according to the Fagerström test | baseline (Day 0), Day 5 (end of iTBS sessions), Day 12 and Day 30 post-iTBS
  Scores achieved on the validated Fagerström scale. The Fagerström test consists of six questions. A score of 0 - 10 is obtained depending on the answers given. A score of 0 - 2 = zero addiction, 3 - 4 = slight addiction, 5 - 6 = moderate addiction, 7 ou 8 heavy addiction and 9 - 10 = very heavy addiction.

CONTACTS AND LOCATIONS:
Overall Officials: Emmanuel HAFFEN, Professor, Principal Investigator — Centre Hospitalier Universitaire de Besancon
Locations (1):
- Magali NICOLIER, Besançon, France

IPD SHARING:
Plan to Share IPD: No